CLINICAL TRIAL: NCT03792828
Title: Pre-emptive Effect of Duloxetine in the Second Knee in Staged Total Knee Arthroplasty: A Randomized Controlled Study
Brief Title: Pre-emptive Effect of Duloxetine in the Second Knee in Staged Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung-Baik Kang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUBMC_20181128
Record Dates: First submitted 2018-11-28; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Knee Osteoarthritis
Keywords: total knee replacement arthroplasty; total knee arthroplasty; central censitization; duloxetine; serotonin-norepinephrine reuptake inhibitors; pre-emptive effect
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Duloxetine HCl 30mg is not used.
  Interventions: Drug: Duloxetine HCl 30mg
- Duloxetine (Experimental): One capsule of Duloxetine HCl 30mg (Duroceptol) is taken orally and daily from the day before the first operation to seven days after the second operation.
  Interventions: Drug: Duloxetine HCl 30mg

INTERVENTIONS:
Drug: Duloxetine HCl 30mg — In the duloxetine group, one capsule of Duloxetine HCl 30mg (Duroceptol) is taken orally and daily from the day before the first operation to seven days after the second operation. In the control group, the patients can take painkillers except duloxetine.

SUMMARY:
In Korea, the interval between knee arthroplasties is usually 1 week. According to previous studies, when total knee arthroplasty was performed at 1-week intervals, total bleeding was reduced and the period of hospital stay was shortened.

However, if stepwise total knee arthroplasty is performed at intervals of one week, the pain is greater after the second operation, and the reason for this phenomenon is known to be due to central sensitization and opioid resistance.

Therefore, the investigators aim to confirm whether Duloxetine reduces the central sensitization as previously known and affects the pain control after the second operation.

DETAILED DESCRIPTION:
Degenerative arthritis of the knee is one of the most common arthritis. Currently, total knee arthroplasty is the most commonly used surgical procedure. The degenerative changes of the knee are often seen on both sides, and bilateral total knee arthroplasty is usually performed. In the past, bilateral total knee arthroplasty was performed at the same time. When bilateral total knee arthroplasty was performed simultaneously, the complications such as increased mortality occurred. So, it is common to perform bilateral total knee arthroplasty in a stepwise manner.

In Korea, the interval between knee arthroplasties is usually 1 week. According to previous studies, when total knee arthroplasty was performed at 1-week intervals, total blood loss was reduced and the period of hospital stay was shortened. However, if stepwise total knee arthroplasty is performed at intervals of one week, the pain is greater after the second operation, and the reason for this phenomenon is known to be due to central sensitization and opioid resistance.

Therefore, the investigators aim to 1) whether the pain is greater than the first operation at the second operation in the control group. 2) whether the pre-operative and post-operative duloxetine use causes the pre-analgesic effect on the second operation. 3) whether the central sensitization, clinical score, and painkiller usage are different by comparing duloxetine-treated group and control group.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for staged bilateral total knee replacement arthroplasty due to osteoarthritis of the knee.

Exclusion Criteria:

* Known allergic reaction to duloxetine
* Secondary arthritis (ex. Rheumatic arthritis, traumatic arthritis, septic arthritis)
* History of major operation(ex. Arthroscopic knee arthroplasty, osteotomy, open reduction, and internal fixation)
* History of manic or bipolar disorder, epilepsy, increased intraocular pressure or risk of acute angle-closure glaucoma, liver disease, moderate renal disease (CLcr < 30ml/min), severe heart disease, uncontrolled hypertension, unregulated narrow-angle glaucoma
* Known congenital or acquired coagulopathy
* Known genetic disorders such as fulminant intolerance / glucose-galactose uptake disorder/sucrose isoleucetase deficiency
* Taken MAO inhibitor, anti-depressants, diuretics, duloxetine
* Refuse to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pain VAS | day 7 (inpatient)
  Pain VAS(11-point numeric scale: 0-11) at rest, maximal knee flexion and maximal knee extension

SECONDARY OUTCOMES:
Central censitization | Preop. day 1, 2, 7 (inpatient) , Postop. 6 week, 3 month
  DN4 (Douleur Neuropathique 4)
Opioid consumption | Preop. day 1, 2, 7 (inpatient) , Postop. 6 week, 3 month
  Opioid conversion to Morphine IV
Pain VAS | Preop. day 1, 2 (inpatient) , Postop. 6 week, 3 month
  Pain VAS(11-point numeric scale: 0-11) at rest, maximal knee flexion and maximal knee extension

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Baik Kang, MD, PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Shin HJ, Kim EY, Na HS, Kim TK, Kim MH, Do SH. Magnesium sulphate attenuates acute postoperative pain and increased pain intensity after surgical injury in staged bilateral total knee arthroplasty: a randomized, double-blinded, placebo-controlled trial. Br J Anaesth. 2016 Oct;117(4):497-503. doi: 10.1093/bja/aew227. Epub 2016 Oct 17. PMID 28077538
- [Background] Scott CE, Murray RC, MacDonald DJ, Biant LC. Staged bilateral total knee replacement: changes in expectations and outcomes between the first and second operations. Bone Joint J. 2014 Jun;96-B(6):752-8. doi: 10.1302/0301-620X.96B6.32793. PMID 24891574
- [Background] Hussain N, Chien T, Hussain F, Bookwala A, Simunovic N, Shetty V, Bhandari M. Simultaneous versus staged bilateral total knee arthroplasty: a meta-analysis evaluating mortality, peri-operative complications and infection rates. HSS J. 2013 Feb;9(1):50-9. doi: 10.1007/s11420-012-9315-7. Epub 2013 Jan 24. PMID 24426845
- [Background] Sun J, Li L, Yuan S, Zhou Y. Analysis of Early Postoperative Pain in the First and Second Knee in Staged Bilateral Total Knee Arthroplasty: A Retrospective Controlled Study. PLoS One. 2015 Jun 11;10(6):e0129973. doi: 10.1371/journal.pone.0129973. eCollection 2015. PMID 26068371
- [Background] Kumar V, Bin Abd Razak HR, Chong HC, Tan AH. Functional Outcomes of the Second Surgery Are Similar to the First in Asians Undergoing Staged-Bilateral Total Knee Arthroplasty. Ann Acad Med Singap. 2015 Nov;44(11):514-8. PMID 27089957
- [Background] Onutu AH. Duloxetine, an antidepressant with analgesic properties - a preliminary analysis. Rom J Anaesth Intensive Care. 2015 Oct;22(2):123-128. PMID 28913467
- [Background] Forster MC, Bauze AJ, Bailie AG, Falworth MS, Oakeshott RD. A retrospective comparative study of bilateral total knee replacement staged at a one-week interval. J Bone Joint Surg Br. 2006 Aug;88(8):1006-10. doi: 10.1302/0301-620X.88B8.17862. PMID 16877597
- [Background] Kim MH, Nahm FS, Kim TK, Chang MJ, Do SH. Comparison of postoperative pain in the first and second knee in staged bilateral total knee arthroplasty: clinical evidence of enhanced pain sensitivity after surgical injury. Pain. 2014 Jan;155(1):22-27. doi: 10.1016/j.pain.2013.08.027. Epub 2013 Aug 30. PMID 23994101
- [Background] YaDeau JT, Brummett CM, Mayman DJ, Lin Y, Goytizolo EA, Padgett DE, Alexiades MM, Kahn RL, Jules-Elysee KM, Fields KG, Goon AK, Gadulov Y, Westrich G. Duloxetine and Subacute Pain after Knee Arthroplasty when Added to a Multimodal Analgesic Regimen: A Randomized, Placebo-controlled, Triple-blinded Trial. Anesthesiology. 2016 Sep;125(3):561-72. doi: 10.1097/ALN.0000000000001228. PMID 27387351